CLINICAL TRIAL: NCT04075617
Title: Cessation of Thumb/Finger Sucking Habit in Children Using Electronic Habit Reminder Versus Palatal Crib.Randomized Clinical Pilot Study.
Brief Title: Cessation of Thumb/ Finger Sucking Habit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tassneim Ahmed, B.D.S, Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Electronic habit reminder
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Thumb/Finger Sucking Habit

STUDY DESIGN:
Masking Description: Blinding isn't feasible except for the statistician.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): electronic habit reminder will fabricated to treat thumb/finger sucking habit containing two parts: acrylic part specially fabricated for the child finger/thumb connected to the reminder in the shape of wrist watch.
  Interventions: Device: electronic habit reminder
- control group (Active Comparator): palatal crib will be cemented after impression taking and fabrication
  Interventions: Other: palatal crib

INTERVENTIONS:
Device: electronic habit reminder — Habit reminder in the form of wrist watch with music that display as reminder is one of recent innovations for cessation of the habit in short time and the child accepts it and it's comfortable
  Arms: intervention group
Other: palatal crib — Fixed palatal crib is commonly used and recommended for treating thumb/finger sucking habit.
  Arms: control group

SUMMARY:
The aim of this study is to assess the use of electronic habit reminder and palatal crib in the cessation of thumb/finger sucking habit.

Treatment of thumb/finger sucking by extraoral approaches are well accepted by school-age children (Adair, 1999). It was reported in a case study by Krishnappa et al that the use of an extraoral electronic habit reminder is a new method used for cessation of thumb/finger sucking habit in short time and it is more comfortable and acceptable to the child (Krishnappa et al, 2016).

DETAILED DESCRIPTION:
This study will be conducted in, Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University. Diagnosis and patient selection will be at outpatient clinic in the specific days of diagnosis. Impression taking, delivery of appliances and follow up will be at post graduate clinic under supervision of the main and assistant supervisor.

Eligible patients will be randomized to form two groups, Intervention group: Treatment by using electronic habit reminder which will be constructed by taking impression for the thumb/finger using silicon impression material (putty consistency) and pouring it with dental stone. The replica of the finger is used to formulate a custom made cover for it, which consists of stainless steel wires with specific design and acrylic resin this is the first part of the reminder. The second part is in the shape of wrist watch which is connected to the first part by a wire. When the child puts his finger in his mouth the stainless steel wires touch each other and the watch produces alarming sound and counts how many times the alarm goes off. The child should wear the appliance most of the time except during eating and activities.

Control group: Treatment by using palatal crib which will be constructed by taking impression for upper arch with alginate impression material, and then will be sent to the lab for fabrication. Cementation of the appliance and then follow up.

Follow up will be at two weeks and 1, 3, 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Children with thumb/finger sucking habit.
* After eruption of upper first permanent molar
* open bite

Exclusion Criteria:

* Patients with special health care need
* Uncooperative child
* Parents refuse the participation of their child

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Cessation of thumb/finger sucking habit | 6 monthes
  cessation of thumb/finger sucking habit is by asking the parent in every appointment during the follow up period if the notice that their child has stopped the habit or at least there is decrease in the duration

SECONDARY OUTCOMES:
child acceptance | 6 monthes
  Child acceptance is simply by asking the child if he/she comfortable/happy with the appliance. The answer is by yes/no
parental acceptance | 6 monthes
  Parental acceptance, there is a questionnaire will be handed to the parent at the end of the treatment period to assess if they found that the device was easy to use, instructions was helpful, the appliance helped in the cessation of the habit and if they will recommend it to others all these questions will be answered by scale (very/somewhat/neutral /minimally/not).And the parents can list if there were any problems they faced with the appliance
time for habit cessation | 6 monthes
  Time for habit cessation is assessed by a booklet is handed to the parent at the beginning of the treatment to record the daily thumb/finger habit activity of the child

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Korany, Lecturer, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Only characters of the children thumb/finger sucking habit will be shared and the result and problems faced during the study

REFERENCES:
- [Background] Adair SM. The Ace Bandage approach to digit-sucking habits. Pediatr Dent. 1999 Nov-Dec;21(7):451-3. PMID 10633521
- [Background] Barber; T.K. and Luke, L. . (1985) Pediatric Dentistry.
- [Background] Dean, J. A. (2016) 'Chapter 22 - Managing the Developing Occlusion', in Dean, J. A. (ed.) McDonald and Avery's Dentistry for the Child and Adolescent (Tenth Edition). Tenth Edit. St. Louis: Mosby, pp. 415-478. doi: https://doi.org/10.1016/B978-0-323-28745-6.00022-3.
- [Background] Farsi, N. M. A. and Pedo, C. (1997) 'Najat M.A. Farsi, BDS, MS Fouad S. Salama BDS, MS, Cert Pedo, DABPD, FAAPD'.
- [Background] Feres MF, Abreu LG, Insabralde NM, de Almeida MR, Flores-Mir C. Effectiveness of open bite correction when managing deleterious oral habits in growing children and adolescents: a systematic review and meta-analysis. Eur J Orthod. 2017 Feb;39(1):31-42. doi: 10.1093/ejo/cjw005. Epub 2016 Feb 3. PMID 26846264
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Insabralde NM, de Almeida RR, Henriques JF, Fernandes TM, Flores-Mir C, de Almeida MR. Dentoskeletal effects produced by removable palatal crib, bonded spurs, and chincup therapy in growing children with anterior open bite. Angle Orthod. 2016 Nov;86(6):969-975. doi: 10.2319/011916-49.1. Epub 2016 May 9. PMID 27159552
- [Background] Krishnappa S, Rani MS, Aariz S. New electronic habit reminder for the management of thumb-sucking habit. J Indian Soc Pedod Prev Dent. 2016 Jul-Sep;34(3):294-7. doi: 10.4103/0970-4388.186750. PMID 27461817
- [Background] Marwah, N. (2018) Textbook of Pediatric Dentistry. Jaypee Brothers,Medical Publishers Pvt. Limited. Available at: https://books.google.com.eg/books?id=ZK52DwAAQBAJ.
- [Background] Paul S. Casamassimo (no date) 'The Thumbgaurd Appliance: Pilot research'. Available at: https://tguard.com/wp-content/uploads/2012/03/southernsmiles.pdf (Accessed: 28 April 2019).
- [Background] Pisani L, Bonaccorso L, Fastuca R, Spena R, Lombardo L, Caprioglio A. Systematic review for orthodontic and orthopedic treatments for anterior open bite in the mixed dentition. Prog Orthod. 2016 Dec;17(1):28. doi: 10.1186/s40510-016-0142-0. Epub 2016 Sep 19. PMID 27615261
- [Background] Severo AL, de Araujo Filho R, Puentes R, Lemos MB, Piluski PF, Lech O. OSTEOID OSTEOMA IN SCAPHOID: CASE REPORT. Rev Bras Ortop. 2015 Nov 4;47(5):656-8. doi: 10.1016/S2255-4971(15)30019-7. eCollection 2012 Sep-Oct. PMID 27047881
- [Background] Shetty RM, Dixit U, Hegde R, Shivprakash PK. RURS' elbow guard: an innovative treatment of the thumb-sucking habit in a child with Hurler's syndrome. J Indian Soc Pedod Prev Dent. 2010 Jul-Sep;28(3):212-8. doi: 10.4103/0970-4388.73796. PMID 21157057
- [Derived] Eltager T, Bardissy AE, Abdelgawad F. Cessation of thumb/finger sucking habit in children using electronic habit reminder versus palatal crib: a randomized clinical pilot study. BMC Oral Health. 2025 Jan 6;25(1):27. doi: 10.1186/s12903-024-05310-6. PMID 39762827